CLINICAL TRIAL: NCT06283251
Title: Pilot Randomized Pediatric RISE (Resource Intervention to Support Equity) Feasibility Study
Brief Title: PediRISE Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other); Children's Cancer Research Fund (Other)
Responsible Party: Principal Investigator, Kira Bona, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-590
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Cancer; Financial Stress; Financial Hardship; Disparities
Keywords: Pediatric Cancer; Financial Stress; Financial Hardship; Disparities
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PediRISE Program Group (Experimental): Participants will be randomized in a 1:1 fashion and will be stratified by site. Participant parents will complete:
  * Baseline survey in-person, by telephone, or virtually.
  * PediRISE program orientation with study team member, in-person or virtual.
  * Optional meeting with certified benefits counselor.
  * Receive fixed funds twice a month for 6 months.
  * Standard supportive care from social worker and/or resource specialist to identify and discuss available resources.
  * End of study survey.
  Interventions: Behavioral: PediRISE Resource Program
- Usual Care Group (No Intervention): Participants will be randomized in a 1:1 fashion and will be stratified by site. Participant parents will complete:
  * Baseline survey in-person, by telephone, or virtually, and orientation with study team member.
  * Standard supportive care from social worker and/or resource specialist to identify and discuss available resources.
  * End of study survey.

INTERVENTIONS:
Behavioral: PediRISE Resource Program — A centrally administered, income-poverty targeted intervention that includes twice-monthly direct provision of unrestricted cash transfers along with benefits counseling to mitigate the risk of loss of means-tested benefits. Funds will be dispersed to families via provided debit card or through personal banking, PayPal, or Venmo.
  Other Names: PediRISE
  Arms: PediRISE Program Group

SUMMARY:
The goal of this research study is to learn whether investigators can successfully give the PediRISE program to families-in other words, whether most families are interested in participating in a study about the PediRISE program, including a 50-50 chance of receiving standard usual care, and a 50-50 chance of receiving the PediRISE support program.

The names of the study groups in this research study are:

* PediRISE Program Group
* Usual Care Group

DETAILED DESCRIPTION:
This is a pilot, multi-center, randomized research study for the feasibility of the administration of the PediRISE program among 40 poverty exposed children with (1) a new diagnosis of childhood cancer at DFCI and Columbia University and among poverty-exposed families with a child with cancer and (2) receiving hematopoietic stem cell transplant (HSCT) at DFCI, Columbia University, or the University of California - San Francisco (UCSF). Randomization means there is an equal chance of being assigned to the PediRISE Program Group or the Usual Care Group.

Study procedures include screening for eligibility, study visits, and completion of surveys and questionnaires.

Participation in this study will last for about 6-months.

It is expected that about 40 pediatric participants with parents/guardians will take part in this research study.

This study is being supported by grants from the American Cancer Society and the Children's Cancer Research Fund.

ELIGIBILITY:
Inclusion Criteria

Cohort 1: Poverty-exposed children with cancer receiving front-line cancer-directed therapy

1. Child diagnosed with de novo cancer
2. Child has established care at a study site and initiated cancer directed therapy in the prior 2-months
3. Child planned to receive at least 4-months of cancer-directed therapy at study site from time of diagnosis per initial cancer treatment plan
4. Child is <18 years at time of enrollment
5. Parent/guardian screened positive for self-reported low-income (<200% FPL)
6. Family primary residence in CA, CT, MA, ME, NH, NJ, NY or RI
7. Provider approval for permission to approach

Cohort 2: Poverty-exposed children with cancer undergoing HSCT

1. Child undergoing allogeneic HSCT for treatment of cancer
2. Child has established care at a study site and is between 30 days prior to start of planned conditioning through day +7 of HSCT at time of enrollment
3. Child planned to receive follow-up care after discharge for HSCT at study site
4. Child is <18 years at the time of enrollment
5. Parent/guardian screen positive for self-reported low-income (<200% FPL)
6. Family primary residence in CA, CT, MA, ME, NH, NJ, NY or RI
7. Provider approval for permission to approach

Exclusion Criteria

Cohort 1: Poverty-exposed children with cancer receiving front-line cancer-directed therapy

1. Planned transfer of child to a non-DFCI or non-Columbia facility for cancer-directed therapy
2. Foreign national family receiving care as an Embassy-pay patient
3. Child is enrolled on embedded correlative health equity aims of open or upcoming clinical drug trials which are powered on descriptive parent-reported poverty data (e.g. AALL1731, DFCI 25-001). Co-enrollment on a poverty intervention study would confound the specified endpoints of these open trial correlative studies
4. Child or household member receiving SSI

Cohort 2: Poverty-exposed children with cancer undergoing HSCT

1. Planned transfer of child to a non-DFCI, non-Columbia, or non UCSF facility for cancer-directed therapy
2. Foreign national family receiving care as an Embassy-pay patient
3. Child is enrolled on embedded correlative health equity aims of open or upcoming clinical drug trials which are powered on descriptive parent-reported poverty data (e.g. AALL1731, DFCI 25-001). Co-enrollment on a poverty intervention study would confound the specified endpoints of these open trial correlative studies
4. Child previously received RISE intervention
5. Child or household member receiving SSI

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant Consent Rate | 1 Day
  The proportion of eligible participants who provide informed consent to participate in the randomized guaranteed income intervention.
Participant Attrition Rate | At 6 months
  The proportion of participants who withdraw from the study, are lost to follow-up, or otherwise do not complete the assigned study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Kira Bona, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Dr. Kira Bona. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1-year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu